CLINICAL TRIAL: NCT03207672
Title: An Open-label Phase 1 Study of E7389 Liposomal Formulation in Subjects With Solid Tumor
Brief Title: Study of E7389 Liposomal Formulation in Participants With Solid Tumor
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-J081-114
Record Dates: First submitted 2017-06-19; First posted 2017-07-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor
Keywords: E7389 liposomal formulation; dose escalation; maximum tolerated dose; pharmacokinetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schedule 1: E7389-LF (Experimental): Participants will receive E7389-liposomal formulation (LF) at a starting dose of 1.0 to 2.5 milligrams per meters squared (mg/m^2), administered as an intravenous (IV) infusion on Day 1 of a 21-day cycle (tri-weekly).
  Interventions: Drug: E7389-LF
- Schedule 2: E7389-LF (Experimental): Participants will receive E7389-LF at a starting dose of 1.0 to 1.5 mg/m^2, administered as an IV infusion on Day 1 and Day 15 of a 28-day cycle (bi-weekly).
  Interventions: Drug: E7389-LF

INTERVENTIONS:
Drug: E7389-LF — intravenous infusion

SUMMARY:
The maximum tolerated dose (MTD) of E7389 liposomal formulation (E7389-LF) will be determined in the dose escalation part. Safety, pharmacokinetics (PK) and efficacy will be assessed using treatment regimen evaluated in dose escalation part in participants with breast cancer (up to 3 prior regimens of chemotherapy) in the expansion part 1 and in participants with adenoid cystic carcinoma (ACC), gastric cancer (GC), esophageal cancer (EGC), small cell lung cancer (SCLC) and breast cancer (with no prior regimens of chemotherapy) in the expansion part 2, 3, 4, 5 and 6 respectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants with advanced, nonresectable, or recurrent solid tumor for which no alternative standard therapy or no effective therapy exists
* Expansion-part 1 only: breast cancer with confirmed diagnosis, human epidermal growth factor (HER2) negative (immunohistochemistry [IHC] 0/1+, or fluorescence in situ hybridization [FISH] negative), prior chemotherapy of anthracycline and taxane (unless contraindicated), and up to 3 prior chemotherapy regimens to advanced or metastatic disease Expansion-part 2 only: nonresectable ACC with confirmed diagnosis and one or more prior chemotherapy regimens (unless contraindicated) Expansion-part 3, 4 and 5 only: nonresectable GC, EGC and SCLC with confirmed diagnosis and 2 or more prior chemotherapy regimens (unless contraindicated) (1 or more prior chemotherapy regimens for EGC participant who received combination therapy of platinum and taxane).

Ex-part 6 only: breast cancer with confirmed diagnosis, HER2 negative (IHC 0/1+, or FISH negative) and without prior chemotherapy regimens to advanced or metastatic disease. Participants with triple-negative breast cancer (TNBC) who are PD-L1 negative as assessed by the site or who are medically determined by the investigator(s) to be ineligible for treatment with atezolizumab and other immune-checkpoint inhibitors will be included.

* Life expectancy of greater than or equal to (>=) 12 weeks
* Eastern Cooperative Oncology Group-Performance Status (ECOG-PS) of 0 to 1
* Japanese participants aged >=20 years at the time of informed consent
* All adverse events (AEs) due to previous anti-cancer therapy have either returned to Grade 0 or 1 except for alopecia and Grade 2 peripheral neuropathy
* Adequate washout period before study drug administration:

  * Chemotherapy, hormonal therapy and radiotherapy: 3 weeks or more
  * Any therapy with antibody: 4 weeks or more
  * Any investigational drug or device: 4 weeks or more
  * Blood/platelet transfusion or granulocyte-colony stimulating factor (G-CSF): 2 weeks or more
* Adequate renal function defined as serum creatinine less than (<) 2.0 milligrams per deciliter (mg/dL) or creatinine clearance >=40 milliliters per minute (mL/min) per the Cockcroft and Gault formula
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) >=2,000/millimeters cubed (mm^3) (>=2.0 × 10^3/microliter [µl])
  * Platelets >=100,000/mm^3 (>=100 × 10^9/Liter [L])
  * Hemoglobin >=9.0 grams (g)/dL (Expansion-part only: >=8.5 g/dL)
* Adequate liver function:

  * Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) less than or equal to (<=) 1.5
  * Total bilirubin <=1.5 × upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert's syndrome
  * Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <=3 × ULN (<=5.0 times ULN in the participants with liver metastases)
* Expansion-part only: At least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Willing and able to give informed consent and comply with all aspects of the protocol

Exclusion Criteria:

* Any of cardiac conditions as follows:

  * Heart failure New York Heart Association (NYHA) Class II or above
  * Unstable ischaemic heart disease (myocardial infarction within 6 months prior to starting study drug, or angina requiring use of nitrates more than once weekly)
  * Prolongation of Fridericia's corrected QT (QTcF) interval to greater than (>) 480 milliseconds (msec)
* History of hypersensitivity reaction by liposomal formulation agent
* Major surgery within 21 days prior to starting study drug
* Previous treatment with eribulin
* Previous radiation therapy encompassing an extensive region including the bone marrow (example, >30% of bone marrow)
* Known intolerance to the study drug or any of the excipients
* Known to be human immunodeficiency virus (HIV) positive
* Active viral hepatitis (B or C) as demonstrated by positive serology or requiring treatment
* Diagnosed with meningeal carcinomatosis
* Participants with brain or subdural metastases or invasion are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (example, radiologic) or symptoms of brain metastases must be stable for at least 4 weeks before starting study treatment.
* Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
* Expansion-part only: history of active malignancy (except for primary tumor, or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, carcinoma in-situ of the bladder or cervix, or early stage gastric/colorectal cancer) within the past 24 months prior to the first dose of study drug
* Evidence of clinically significant disease/status (example, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [β-hCG] or hCG test). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Males with impregnate potential or females of childbearing potential who or whose partner do not agree with medically effective method of contraception throughout the entire study period and for 28 days (90 days for male) after study drug discontinuation
* Ex-part 6 only: Active or acute oral infection requiring dental treatment
* Ex-part 6 only: Participants who received taxanes as neoadjuvant or adjuvant chemotherapy and have radiographically progressive disease by investigator(s) decision within 12 months after the last dose of taxane
* Ex-part 6 only: Child-Pugh score B or C

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of E7389 liposomal formulation (E7389-LF) | Cycle 1 (21 days): Schedule 1; Cycle 1 (28 days): Schedule 2
  The MTD is defined as the maximum dose with 0 or 1 dose-limiting toxicity (DLT) in 6 participants. DLTs are defined as study drug-related adverse events (AEs) and graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) 4.03 occurring during Cycle 1 (Schedule 1: 3 weeks; Schedule 2: 4 weeks) of the Dose Escalation part of the study (DE-part).

SECONDARY OUTCOMES:
Number of participants with any serious adverse event (SAE) | From date of first dose of study drug up to 30 days after last administration of study drug (approximately up to 8 years)
  The number of participants with any SAE will be assessed as a measure of the safety and tolerability of E7389- liposomal formulation (LF).
Number of participants with any adverse event (AE) | From date of first dose of study drug up to 30 days after last administration of study drug (approximately up to 8 years)
  The number of participants with any AE will be assessed as a measure of the safety and tolerability of E7389-LF.
Maximum observed concentration (Cmax) of E7389-LF | DE part: predose; 15 minutes (min) after start of infusion (inf); 5 min after end of inf on Cycle 1 Day 1 (C1D1); 0.5, 1, 2, 4, 6, 8, and 24 hours (hr) postdose (from end of inf on C1D1); C1D4; C1D8; C1D10. Exp part: predose and end of inf on C1D1; C1D8
  Blood samples will be collected for pharmacokinetic (PK) analyses. Cmax is the highest concentration of drug in the blood that is measured after a dose. DE = Dose Escalation. Exp = Expansion.
Time from dosing to the maximum observed concentration (Tmax) of E7389-LF | DE part: predose; 15 minutes (min) after start of infusion (inf); 5 min after end of inf on Cycle 1 Day 1 (C1D1); 0.5, 1, 2, 4, 6, 8, and 24 hours (hr) postdose (from end of inf on C1D1); C1D4; C1D8; C1D10. Exp part: predose and end of inf on C1D1; C1D8
  Blood samples will be collected for PK analyses. Tmax is the time to the highest concentration of drug in the blood that is measured after a dose. DE = Dose Escalation. Exp = Expansion.
Area under the plasma concentration time course profile (AUC) | DE part: predose; 15 minutes (min) after infusion (inf) start; 5 min after end of inf on Cycle 1 Day 1 (C1D1); 0.5, 1, 2, 4, 6, 8, and 24 hours (hr) postdose (from end of inf on C1D1); C1D4; C1D8; and C1D10. Exp part: predose and end of inf on C1D1; C1D8
  Blood samples will be collected for PK analyses. AUC represents the overall amount of drug in the bloodstream after dosing. DE = Dose Escalation. Exp = Expansion.
Half-life (t1/2) of E7389-LF | DE part: predose; 15 minutes (min) after start of infusion (inf); 5 min after end of inf on Cycle 1 Day 1 (C1D1); 0.5, 1, 2, 4, 6, 8, and 24 hours (hr) postdose (from end of inf on C1D1); C1D4; C1D8; C1D10. Exp part: predose and end of inf on C1D1; C1D8
  Blood samples will be collected for PK analyses. t1/2 is the time required for the concentration of the drug to reach half of its original value. DE = Dose Escalation. Exp = Expansion.
Clearance (CL) of E7389-LF | DE part: predose; 15 minutes (min) after infusion (inf) start; 5 min after end of inf on Cycle 1 Day 1 (C1D1); 0.5, 1, 2, 4, 6, 8, and 24 hours (hr) postdose (from end of inf on C1D1); C1D4; C1D8; and C1D10. Exp part: predose and end of inf on C1D1; C1D8
  Blood samples will be collected for PK analyses. Clearance is the volume of plasma cleared of the drug per unit time. DE = Dose Escalation. Exp = Expansion.
Volume of distribution (Vd) of E7389-LF | DE part: predose; 15 minutes (min) after infusion (inf) start; 5 min after end of inf on Cycle 1 Day 1 (C1D1); 0.5, 1, 2, 4, 6, 8, and 24 hours (hr) postdose (from end of inf on C1D1); C1D4; C1D8; and C1D10. Exp part: predose and end of inf on C1D1; C1D8
  Blood samples will be collected for PK analyses. Vd is the volume in which a drug is distributed. DE = Dose Escalation. Exp = Expansion.
Objective response rate (ORR) | From date of first dose of study drug until first documentation of CR or PR (up to approximately 8 years)
  ORR is defined as the percentage of participants who have a best overall response of complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. For target lesions, CR is defined as the disappearance of all target lesions. For non-target lesions, CR is defined as the disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (less than [<] 10 millimeter [mm] short axis). Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. For target lesions, PR is defined as at least a 30 percent (%) decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Progression free survival (PFS) | From the date of first dose of study drug until progressive disease (PD), death, whichever occurs first (up to approximately 8 years)
  PFS is defined as the time from the date of first dose of study drug to the date of the first documentation of disease progression or date of death, whichever occurs first. For target lesions PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, progressive disease is defined as the unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.

CONTACTS AND LOCATIONS:
Locations (12):
- Japan (12):
  - Eisai Trial Site 3, Kashiwa, Chiba
  - Eisai Trial Site 5, Sapporo, Hokkaido
  - Eisai Trial Site 8, Nishinomiya, Hyōgo
  - Eisai Trial Site 6, Yokohama, Kanagawa
  - Eisai Trial Site 10, Hidaka, Saitama
  - Eisai Trial Site 9, Bunkyo-ku, Tokyo
  - Eisai Trial Site 1, Chuo-ku, Tokyo
  - Eisai Trial Site 4, Koto-ku, Tokyo
  - Eisai Trial Site 7, Shinjuku-ku, Tokyo
  - Eisai Trial Site 12, Fukuoka
  - Eisai Trial Site 11, Kyoto
  - Eisai Trial Site 2, Osaka

REFERENCES:
- [Derived] Masuda N, Ono M, Mukohara T, Yasojima H, Shimoi T, Kobayashi K, Harano K, Mizutani M, Tanioka M, Takahashi S, Kogawa T, Suzuki T, Okumura S, Takase T, Nagai R, Semba T, Zhao ZM, Ren M, Yonemori K. Phase 1 study of the liposomal formulation of eribulin (E7389-LF): Results from the breast cancer expansion cohort. Eur J Cancer. 2022 Jun;168:108-118. doi: 10.1016/j.ejca.2022.03.004. Epub 2022 Apr 29. PMID 35500404
- [Derived] Sato J, Shimizu T, Koyama T, Iwasa S, Shimomura A, Kondo S, Kitano S, Yonemori K, Fujiwara Y, Tamura K, Suzuki T, Takase T, Nagai R, Yamaguchi K, Semba T, Zhao ZM, Ren M, Yamamoto N. Dose Escalation Data from the Phase 1 Study of the Liposomal Formulation of Eribulin (E7389-LF) in Japanese Patients with Advanced Solid Tumors. Clin Cancer Res. 2022 May 2;28(9):1783-1791. doi: 10.1158/1078-0432.CCR-21-3518. PMID 35180771